CLINICAL TRIAL: NCT03868605
Title: Endoscopic Full Thickness Resection Versus Standard Therapy of the Colorectal Neoplasia - Prospective Randomized Study
Brief Title: Endoscopic Full Thickness Resection Versus Standard Therapy of the Colorectal Neoplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Collaborators: Masaryk University (Other); University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Stepan Suchanek, MD., Ph.D., Head of Endoscopy unit, Military University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-18-08-00246
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Polyps; Colon Cancer
MeSH Terms: conditions — Polyps; Colonic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMR/ESD (Experimental): Standard EMR or ESD technique
  Interventions: Device: EMR and ESD
- Over- the- scope full- thickness resection device (Experimental): Endoscopic full thickness resection
  Interventions: Device: Over- the- scope full- thickness resection device

INTERVENTIONS:
Device: EMR and ESD — Endoscopic mucosal resection using a resection snare Endoscopic submucosal dissection using an electrosurgical knife
  Arms: EMR/ESD
Device: Over- the- scope full- thickness resection device — Endoscopic resection of neoplastic lesions of the colon using the over- the- scope full- thickness resection device
  Arms: Over- the- scope full- thickness resection device

SUMMARY:
Most of the cancers develop from the adenomatous polyps. The therapeutic methods have been established already - endoscopic polypectomy (EPE) for stalked polyps and endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) for non-pedunculated polyps. EMR is preferred in European countries over ESD because of its higher feasibility. However, the local residual neoplasia (LRN) after EMR has been reported in 14 - 24 % cases. There is a higher LRN risk in sessile polyps which do not elevate sufficiently after the submucosal injection (non-lifting sign) and the piece-meal resection needs to be used. Therefore, the new method of endoscopic full-thickness resection (FTR) has been developed to resect these lesions.

DETAILED DESCRIPTION:
In this project, 80 individuals (age ≥ 18 years) with colorectal lesions of 10-25 mm size with positive non-lifting sign will be included. Such lesions might be found during the colonoscopies at the trial endoscopy centers or at the cooperating referring endoscopy centers outside the study. Patient will be scheduled for the index therapeutic colonoscopy (iTC) and randomized in two groups - FTR group (therapy with FTRD) and ST group (standard therapy, EMR or ESD due to the indication, decided by the endoscopist). First follow-up colonoscopy (FC1) will be performed in 6 months interval. In case of LRN negativity at FC1, the second follow-up colonoscopy (FC2) will be done after 12 months (18 months since iTC). In case of LRN positivity at FC1, the LRN therapeutic colonoscopy (LRN-TC) will follow with the endoscopic method due the findings (patients will be divided into four groups): APC group (LRN ≤ 5 mm; APC therapy), EMR group (LRN > 5 mm and negative non-lifting sign negative; EMR therapy), FTR group (LRN > 5 mm and positive non-lifting sign; therapy with FTRD) and surgery group (complex lesion; surgical therapy). In some LRN positive cases, FC1 will be the same as LRN-TC. The first follow-up colonoscopy after LRN therapy (LRN-FC1) will be performed after 6 months (12 months since TC). In case of re-LRN negativity at LRN-FC1 the second follow-up colonoscopy after LRN therapy (LRN-FC2) will be done after 6 months (18 months since iTC). In case of re-LRN positivity at LRN- FC1 the therapy will be done same as during FC1 and next follow-up will be done outside this trial. In some re-LRN positive cases, LRN-FC1 will be the same as re-LRN-TC. In conclusion, all patients will be followed-up within the study for 18 months, if timely possible.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* colorectal lesions of 10-25 mm size with positive non-lifting sign
* signed informed consent with the study and with colonoscopy

Exclusion Criteria:

* age < 18 years
* lesions > 25 mm
* pedunculated polyps
* colorectal stenosis
* colonoscopy contraindication
* severe acute inflammatory bowel disease
* severe comorbidities
* patient not able to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of R0 procedures | 3 months
  proportion of patients with resection specimens with negative horizontal and vertical margins confirmed by histopathology

SECONDARY OUTCOMES:
Proportion of curative resections | 12 months
  Proportion of the LRN at 6 months and 12 months follow-up colonoscopy after the index therapeutic colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Suchanek, MD., Ph.D, Principal Investigator — Military University Hospital, Prague
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided